CLINICAL TRIAL: NCT06490380
Title: A Collaborative Project Aimed to Establish a WGS-based Reference Standard for Evaluating the Analytical Performance of HRD Status Testing
Brief Title: HRD Status Reference Standard Based on WGS
Status: Completed | Type: Observational
Sponsor: Lei Li (Other)
Collaborators: National Institutes for Food and Drug Control, China (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: HRDref-WGS
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PARPi — Poly(adenosine diphosphate-ribose) polymerase inhibitor (PARPi)

SUMMARY:
When evaluating the analytical performance of homologous recombination deficiency (HRD) status testing, there is currently no widely accepted reference standard. Therefore, a collaborative project was initiated to establish a HRD status reference standard for the industry. Although there is no genotyping strategy that is universally recognized as the most accurate for evaluating HRD status, whole-genome sequencing (WGS) is one of the best candidates.

DETAILED DESCRIPTION:
* Primary objective: To establish a HRD status reference standard based on WGS.
* Secondary objective: To validate the analytical performance of panel HRD status using WGS HRD status as reference standard.
* Exploratory objective 1: To explore how methylation of selective genes correlate with WGS HRD status and efficacy.
* Exploratory objective 2: To explore how HRR gene mutations correlate with WGS HRD status and efficacy.
* Exploratory objective 3: To set up a harmonized bioinformatic analysis workflow for WGS HRD status.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at diagnosis
* Ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
* High-grade serous or high-grade endometroid histological type
* FIGO stage II, III, or IV
* Complete response or partial response following completion of first-line adjuvant chemotherapy
* PARPi administered as first-line maintenance therapy

Exclusion Criteria:

* First-line surgery not conducted
* Total round of first-line chemotherapy (neoadjuvant and adjuvant) less than 5
* First-line PARPi maintenance therapy initiated beyond 12 weeks after last dose of chemotherapy
* Genotyping quality-control failed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer patients received first-line PARPi maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to 42 months
  Time from first dose of PARPi to disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | Up to 48 months
  Time from first dose of PARPi to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No